CLINICAL TRIAL: NCT02270229
Title: Evaluation of the Peritoneal Dialysis Program in a Hospital in Chinandega, Nicaragua.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: La Isla Foundation (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: rev5162014
Record Dates: First submitted 2014-09-29; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Kidney Disease; Peritoneal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (4):
- Healthcare providers
- PD patients
- Primary caregivers of the PD patients
- Laboratory personnel

SUMMARY:
The purpose of this study is to develop recommendations to assist in improving the current peritoneal dialysis (PD) program in a Hospital in Chinandega, Nicaragua. This project will consist of a needs assessment, a review of aggregate quantitative patient data from hospital records, and a knowledge, attitudes, and practices (KAP) assessment for medical providers, laboratory technicians, patients and primary caregivers. The final report will be used to obtain funding for the implementation of the recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be affiliated with the PD program that is under evaluation

Exclusion Criteria:

1. Being physically unable to participate in an interview of approximately one hour
2. Being younger than 18 years of age
3. Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed in a public hospital in northwest Nicaragua.
  There will be four groups of participants:
  1. Healthcare professionals, including physicians, nurses, technicians, and administrators
  2. PD patients
  3. Primary caregivers of the PD patients
  4. Laboratory personnel
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Identification of needs of the PD program | Hospital visits for the duration of 1 week
  This outcome will be measured by filling out a pre-designed checklist based on national and international guidelines, including equipment, material and staffing needs.
Adherence to established protocols on administering PD treatment in the hospital | 3 days of observation sessions for the duration of 8 hours
  This outcome will be measured by filling out a validated checklist of steps that need to be performed by the healthcare provider while PD is administered in the Hospital
Levels of knowledge, attitudes and practices towards PD of healthcare providers, laboratory staff patients and primary caregivers | Interviews of each group for the duration of 1 week
  This outcome will be measured by administering a questionnaire to the participants of 4 respective groups (healthcare providers, laboratory staff, patients, primary caregivers). The questionnaire will contain sections on (1) demographic information/professional affiliation with the program, (2) knowledge of PD, (3) attitudes towards PD, (4) practices regarding PD, and (5) perceived needs of the program. The levels of knowledge will be classified in four categories: 1) very good, 2) good, 3) regular, 4) poor. Attitudes will be classified as either positive or negative. Practices will be classified as either good or bad.
Prevalence of peritonitis and causative agents | Sample collections according to PD patients' appointment times during one week and culturing of samples for 72 hours
  This outcome will be measured by identifying pathogens in patients' dialysate liquid and estimating the overall percentage of patients with peritonitis.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Gonzalez, MD. MSc., Principal Investigator — CISTA UNAN-Leon